CLINICAL TRIAL: NCT05377892
Title: Modulating Dietary Protein to Alter Circulating and Gut Metabolites
Brief Title: The Impact of Dietary Protein on the Metabolome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, David Montrose, Assistant Professor, Pathology, Stony Brook University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: IRB2019-00415
Record Dates: First submitted 2022-05-04; First posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Diet, Healthy
MeSH Terms: interventions — Dietary Proteins

STUDY DESIGN:
Intervention Model Description: Longitudinal
Masking Description: single blinded (participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Subjects receiving high protein followed by reduced protein diet
  Interventions: Other: Dietary protein

INTERVENTIONS:
Other: Dietary protein — High protein followed by reduced protein diet

SUMMARY:
It is known that tumors have an affinity for taking up amino acids from circulation or nearby tissues to use as a fuel source, to enhance their growth. Work in rodents has shown that when the levels of amino acids are reduced in diet, tumor growth is slowed and tumors are more susceptible to anti-cancer therapies. There are limited evidence-based dietary recommendations for cancer patients, which represents an urgent and unmet need. It is likely that reducing dietary protein will be beneficial, however this has not been tested. In advance of carrying out a study in cancer patients a study in healthy volunteers needs to be conducted to determine whether altering the amount of dietary protein, impacts the levels of amino acids (or other metabolites) in blood or the intestine. By demonstrating that altering dietary protein can alter the metabolome of healthy individuals, it will provide the information needed to reduce protein intake in cancer patients in future studies.

DETAILED DESCRIPTION:
After providing consent, subjects will undergo an indirect calorimetry test, which involves breathing through a disposable, single-use mouth piece into a machine that estimates calorie needs based on oxygen consumed and CO2 produced. Then subjects will be instructed on how to keep a 3-day food record and complete the Qualtrics survey designed for this purpose within 2 weeks of consenting. Nutrient content of the participants' typical diet will be calculated, based on the 3-day and Qualtrics-based food/beverage log, using Food Processor software. Meals for the acclimation period will be created to mimic the participants' typical diet (daily calories and percent of calories from carbohydrate, protein and fat), as well as to meet their calorie needs per the indirect calorimeter test, for the first 7-9 days of the study. High protein diets (2g of protein/kg/day) will then be devised and provided for the next 14-16 days. Following this period, reduced protein diets (0.8g of protein/kg/day) will be devised and provided for the next 14-16 days. Fat content will be modulated to keep diets isocaloric while keeping carbohydrate content stable. Participants will choose between two 3-day cycle menus for each feeding phase. Meals will be prepared in a metabolic kitchen housed in SBU's Business Incubator at Calverton. Meals will be prepared in batches, packaged and frozen at the incubator, then transported in a cooler with thermometers to the Food Service Department at SBU Hospital. Meals will be kept frozen in freezers until the day they are provided to participants. Logs of temperatures of coolers will be maintained daily, with temperatures checked every hour.

In order to provide meals, participants will come to the feeding site to eat breakfast onsite and pick up other meals and snacks for the rest of the day. Participants will be provided a closed envelope containing a form that will list their participant ID# and age in which they'll sign in and indicate if they've begun any new medications or been diagnosed with a disease since starting the study. Additionally, twice per week, participants will be weighed using a digital scale in order to track changes in body weight while on the study. If weight changes greater than 2% of baseline, calorie content of the meals will be modified to avoid further weight changes. Food for the rest of the day will be provided in an insulated bag containing frozen cold packs and participants will be instructed to keep lunch and dinner in the insulated bag or a refrigerator until eaten. They will be instructed to heat the respective meals in a microwave until hot, prior to consumption. They will be instructed to take a picture of each meal before and after eating and upload the pictures via a Qualtrics-based survey, in order for the investigators to estimate how much food has been eaten at each meal. Although participants will be instructed to only eat the food and beverages provided for the study, they will log any consumption of food or beverages not provided for the study via this same Qualtrics-based survey. Consumption of water, black coffee and tea will not be logged.

During days 7-9, 24-26 and 41-43 participants will provide a stool sample to be placed into a sterile container (provided by the study team) then placed into an opaque brown paper bag and provided to the study team. At the same time the stool sample is delivered, blood will be drawn to generate serum. If a participant provides samples in the earlier part of the collection period (e.g. day 7) they will proceed immediately to the next phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30 years
* BMI 18-29.9

Exclusion Criteria:

* Those with a history of significant illness including diabetes, renal, liver or cardiovascular disease, malnutrition, GI disease (including IBS, IBD, chronic constipation or diarrhea), mental illness (i.e. depression, bipolar disorder)
* Those adhering to a vegetarian or vegan diet.
* Those having taken antibiotics within 1 month of starting the study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 9 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Subject reported adherence to study diet. | 5 weeks
  Participants will take a picture of each meal before and after eating and upload the pictures via a Qualtrics-based survey. The investigators will use these images to estimate how much food has been eaten at each meal, then calculate macronutrient intake based on the nutrient content of each food item. Participants will log any consumption of food or beverages not provided for the study via this same Qualtrics-based survey in order to estimate the contribution of non-study foods to overall macronutrient consumption. The average percent change in protein intake across subjects after switching from acclimation to high protein or high protein to reduced protein stages will be quantified.
Mass spectrometry-based measurement of abundance of metabolites in blood | 4 weeks
  Global metabolite profiling will be carried out using mass spectrometry on blood collected at the end of the acclimation, high protein and reduced protein stages. Data will be log transformed and paired t tests will be conducted to determine if significant changes in abundance occur following consumption of high protein or reduced protein diets
Mass spectrometry-based measurement of abundance of metabolites in stool | 4 weeks
  Global metabolite profiling will be carried out using mass spectrometry on stool collected at the end of the acclimation, high protein and reduced protein stages. Data will be log transformed and paired t tests will be conducted to determine if significant changes in abundance occur following consumption of high protein or reduced protein diets

CONTACTS AND LOCATIONS:
Overall Officials: David Montrose, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
publication of results in scientific journal
Supporting Information: Study Protocol, SAP
Time Frame: 2022; indefinitely
Access Criteria: subscription access to journal

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-23): https://cdn.clinicaltrials.gov/large-docs/92/NCT05377892/Prot_SAP_000.pdf